CLINICAL TRIAL: NCT03336047
Title: The Effect of Personal Activity Intelligence Versus 10,000 Steps Daily on Cardiorespiratory Fitness in Overweight and Obese
Brief Title: The Effect of Personal Activity Intelligence Versus 10,000 Steps Daily on Cardiorespiratory Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1211
Record Dates: First submitted 2017-11-01; First posted 2017-11-08 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Obesity; Physical Activity
Keywords: Exercise; Actigraphy; Prevention and Control; Cardiorespiratory Fitness
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10,000 steps daily (Active Comparator): Subjects will be encouraged to obtain 10 000 steps a day, monitored by a step counter (fit bit zip)
  Interventions: Behavioral: 10,000 steps daily
- using personal activity intelligence (Experimental): Subjects will be encouraged to obtain 100 PAI points per week, monitored by Mio Slice and the Mio Pai 2.0 smart phone application
  Interventions: Behavioral: personal activity intelligence

INTERVENTIONS:
Behavioral: personal activity intelligence — Participants randomized to the PAI intervention will receive a Mio Slice fitness bracelet and asked to install the Mio Pai 2.0 app on their smart phone. This tracks their fitness score based on the PAI algorithm where the goal is to maintain 100 PAI points a week. PAI is earned incrementally based on time spent in three different heart rate zones, low, medium and high intensity. PAI is recorded every day and added to the weekly total and the PAI earned on the same day the previous week is deleted (on Tuesday, the PAI earned the previous Tuesday will disappear).
  Participants will be encouraged to maintain 100 PAI during the 8 weeks intervention by telephone messages (sms).
  Other Names: PAI
  Arms: using personal activity intelligence
Behavioral: 10,000 steps daily — Participants randomized to the 10,000 step intervention will receive a fit bit zip step counter and asked to obtain 10.000 steps per day. Participants will be encouraged to obtain 10.000 steps per day by telephone messages (sms).
  Arms: 10,000 steps daily

SUMMARY:
A high physical fitness can prevent cardiovascular disease. Which form of exercise training is efficient at improving fitness is well known. The challenge is to get people to do it. Personal activity intelligence (PAI) is an algorithm developed for this challenge. It gives a score that tells the users whether they are active enough to achieve the maximum health benefit of exercise based on their heart rate. It has been shown that people who obtain 100 PAI a week have less cardiovascular disease, but intervention studies showing that PAI can improve physical fitness are so far lacking.

Step counters have received a lot of attention and 10 000 steps a day is a common recommendation, but little is known about the physiological adaptations to this intervention.

This study will compare the effect of physical activity with a value of 100 PAI points a week with 10 000 steps a day in healthy, but overweight (body mass index > 25) participants between 30 and 50 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 25
* Low physical activity (less than 50 PAI points calculated from a questionnaire)

Exclusion Criteria:

* Cancer diagnosis
* Cardiac arrhythmia
* Angina
* Previous myocardial infarction
* lung disease
* heart disease
* uncontrolled hypertension
* kidney disease
* orthopedic or neurological limitations
* planned surgery during the intervention
* participation in other research studies conflicting with the current study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | After the intervention period (8 weeks)
  The highest amount of oxygen the body can take up, achieved at maximal exercise at the end of an incremental treadmill test measured through ergospirometry. The difference between the two groups post-intervention will be used, while controlling for a pre-intervention value.

SECONDARY OUTCOMES:
Body composition | After intervention period (8 weeks)
  Body mass, fat mass and lean mass will be measured using a bio impedance analysis which weighs the participants and uses bio impedance to also assess fat mass and lean mass.
  The difference between the two groups post-intervention will be used, while controlling for a pre-intervention value.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Hjulstad Bækkerud, Principal Investigator — Norwegian University of Science and Technology; Ulrik Wisløff, phd prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Trondheim, Sør Trøndelag, Norway